CLINICAL TRIAL: NCT05133921
Title: The Clinical Efficacy and Safety of Drug-coated Balloon in Coronary Lesions: a Real-World, All-Comers ,Single-center, Prospective Study
Brief Title: The Clinical Efficacy and Safety of Drug-coated Balloon
Status: Completed | Type: Observational
Sponsor: Xijing Hospital (Other)
Responsible Party: Principal Investigator, Ling Tao, MD, PhD, Professor in Cardiology, Director of the department of Cardiology, Xijing Hospital
Other Study IDs: CAGE-FREE registry
Record Dates: First submitted 2021-11-22; First posted 2021-11-24 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-02

CONDITIONS: Coronary Heart Disease; Angioplasty, Balloon
Keywords: Drug-coated balloons; De-novo; All-comers; In-stent stenosis
MeSH Terms: conditions — Coronary Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Drug-Coated Balloon (DCB) angioplasty is similar to plain old balloon angioplasty procedurally, but there is an anti-proliferative medication paclitaxel coated on the balloon. Treating in-stent restenosis (ISR) with the DCB has the theoretical advantage of avoiding multiple stent layers and respecting the vessel anatomy. DCB has shown promising results for the treatment of ISR. Currently, DCB has a Class I indication to treat ISR recommended by European Society of Cardiology (ESC) guidelines. In addition, some interventional cardiologist has also applied DCB in de novo lesions in their clinical practice.

Although some small sample size RCTs and observational studies have suggested that the clinical prognosis of DCB in primary large vessels is non-inferior to drug-eluting stent (DES), there is no large-scale RCT or cohort studies to compare the clinical effects of DCB and DES.

Despite several theoretical benefits of DCB, the procedural-related complications cannot be entirely prevented, such as acute elastic retraction and severe dissection, which would affect coronary blood flow or lead to acute vascular occlusion.

Some studies have suggested that optimization of the procedural technique can reduce the occurrence of complications and target lesion failure in the long-term. Proposed criteria include adapting cutting or scoring balloon for pre-dilatation, residual stenosis<30% post-DCB, maintaining TIMI flow=3, DCB dilation time<60s, and appropriate balloon to vessel ratio> 0.91. However, such proposed technique and criteria have not been evaluated in the real-world clinical practice.

This current study is designed to investigate the efficacy and safety of DCB in the real world and exploring the optimal procedural configurations.

ELIGIBILITY:
Inclusion Criteria:

1. Patients who received PCI with one or more drug-coated balloons (DCB)
2. Patients who did not received drug-eluting stent implantation

Exclusion Criteria:

1. Currently participating in another trial or participants unable to comply to follow-up

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All patients who received PCI with one or more drug-coated balloons (DCB) in the Xijing hospital of the Air Force Medical University from December 1, 2015 to December 1, 2019.
Sampling Method: Non-Probability Sample
Enrollment: 2487 (Actual)
Dates: Start 2015-12-01 (Actual); Primary Completion 2020-12-01 (Actual); Study Completion 2020-12-01 (Actual)

PRIMARY OUTCOMES:
Device-oriented Composite Endpoint (DoCE) | 24 months
  DoCE is a composite clinical endpoint of cardiac death, target vessel myocardial infraction (TV-MI), and Clinically individual target lesion revascularization (CI-TLR)

OTHER OUTCOMES:
Device-oriented Composite Endpoint (DoCE) | 1 month, 1, 2, 3, 5, 7, 10 years
  DoCE is a composite clinical endpoint of cardiac death, target vessel myocardial infraction (TV-MI), and Clinically individual target lesion revascularization (CI-TLR)
POCE | 1 month, 1, 2, 3, 5, 7, 10 years
  POCE is a composite clinical endpoint of all-cause death, any stroke, non-fatal myocardial infarction (MI), any revascularization
All-cause death | 1 month, 1, 2, 3, 5, 7, 10 years
  Rates of individual components of PoCE
Non-fatal myocardial infarction (MI) | 1 month, 1, 2, 3, 5, 7, 10 years
  Rates of individual components of PoCE
Any stroke | 1 month, 1, 2, 3, 5, 7, 10 years
  Rates of individual components of PoCE
Any revascularization | 1 month, 1, 2, 3, 5, 7, 10 years
  Rates of individual components of PoCE
Cardiac death | 1 month, 1, 2, 3, 5, 7, 10 years
  Rates of individual components of DoCE
Target vessel myocardial infraction (TV-MI) | 1 month, 1, 2, 3, 5, 7, 10 years
  Rates of individual components of DoCE
Clinically individual target lesion revascularization (CI-TLR) | 1 month, 1, 2, 3, 5, 7, 10 years
  Rates of individual components of DoCE
Target vessel failure (TVF) | 1 month, 1, 2, 3, 5, 7, 10 years
  Target vessel failure is defined as cardiovascular death, target vessel myocardial infraction (TV-MI), and clinically-indicated target vessel revascularization
Clinically-indicated target vessel revascularization | 1 month, 1, 2, 3, 5, 7, 10 years
  Rates of individual components of TVF
BARC type 3 or 5 bleeding events | 1 month, 1, 2, 3, 5, 7, 10 years
  Bleeding events type 3 or 5 defined by BARC (Bleeding Academic Research Consortium) criteria
Net adverse clinical events (NACE) | 1 month, 1, 2, 3, 5, 7, 10 years
  NACE is a composite clinical endpoint of all-cause death, any stroke, any any non-fatal myocardial infarction ( MI) any revascularization and BARC type 3 or 5 bleeding events
Vessel-oriented Composite Endpoint (VOCE) | 1 month, 1, 2, 3, 5, 7, 10 years
  VOCE is a composite clinical endpoint of Vessel-related cardiovascular Death, Target-vessel related MI, Clinically-oriented Target vessel revascularization
Vessel-related cardiovascular Death | 1 month, 1, 2, 3, 5, 7, 10 years
  Rates of individual components of VOCE

CONTACTS AND LOCATIONS:
Overall Officials: Ling Tao, MD, Ph.D., Study Chair — Xijing Hospital; Chao Gao, MD, Ph.D., Study Chair — Xijing Hospital
Locations (1):
- Ling Tao, Xi'an, Shannxi, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] He X, Liu Y, Yin Z, Li F, van Geuns RJ, Garg S, Onuma Y, Serruys PW, Gao C, Tao L. Mid-term outcomes of paclitaxel-coated balloon for de novo non-small coronary lesions: a pooled analysis. BMC Med. 2025 Oct 31;23(1):598. doi: 10.1186/s12916-025-04429-9. PMID 41174582